CLINICAL TRIAL: NCT06396845
Title: Assessing the Benefits of Robotic and Laparoscopic Surgery for Mid and Low Rectal Cancer in Patients: The Charlson Comorbidity Index (CCI)
Status: Completed | Type: Observational
Sponsor: Daorong Wang (Other)
Responsible Party: Sponsor-Investigator, Daorong Wang, DR, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Other Study IDs: CCI1
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Robotic; Laparoscopic; Anterior Resection for Rectal Cancer
MeSH Terms: interventions — Robotic Surgical Procedures; Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- robotic surgery with cci
  Interventions: Procedure: robotic surgery; Procedure: laparoscopic surgery
- laparoscopic surgery with cci
  Interventions: Procedure: robotic surgery; Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: robotic surgery — robotic surgery
Procedure: laparoscopic surgery — laparoscopic surgery

SUMMARY:
This retrospective study collected participants who underwent robotic or laparoscopic anterior resection for rectal cancer at the North People's Hospital in Jiangsu from January 2019 to January 2023.

ELIGIBILITY:
Inclusion Criteria:

The criteria include: (1) pathology of low rectal cancer (within 10 cm from the anal margin); (2) access to comprehensive pathological and computed tomography (CT) data; (3) completeness of clinical data.

Exclusion Criteria:

patients with other malignant tumors besides rectal cancer, benign disease surgery, and emergency surgery.

Ages: 55 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants who underwent robotic or laparoscopic anterior resection for rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
postoperative recurrence rate | 2018-2024
  postoperative recurrence rate

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Jiangsu People's Hospital, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No